CLINICAL TRIAL: NCT03005964
Title: A Multi-Center, Double-Blind, Randomized, Vehicle- Controlled, Parallel-Group Study Comparing AM001 Cream, 7.5% to Vehicle Cream in the Treatment of Plaque Psoriasis
Brief Title: Safety and Efficacy Study Comparing AM001 Cream, 7.5% to Vehicle Cream in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AmDerma (Industry)
Collaborators: International Dermatology Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AD-AM001-001A
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — potassium dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AM001 Cream, 7.5% (Experimental): A white to off-white Cream free from any foreign particles
  Interventions: Drug: AM001 Cream, 7.5%
- Vehicle Cream (Placebo Comparator): A white to off-white Cream free from any foreign particles.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: AM001 Cream, 7.5% — Active Cream
  Other Names: Potassium Dobesilate
  Arms: AM001 Cream, 7.5%
Drug: Vehicle Cream — Placebo
  Other Names: Placebo Cream
  Arms: Vehicle Cream

SUMMARY:
To compare the safety and efficacy profiles of AM001 Cream, 7.5% and its vehicle cream in the treatment of plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent.
2. Subjects must be male or female, at least 18 years of age.
3. Subjects with a definite diagnosis of plaque psoriasis that is clinically active (for at least 3 months), involving at least 10% and up to 20% of the body surface area (not including the head [ scalp, face], hands, feet, and intertriginous areas).
4. Subjects with an Investigator's Global Assessment (IGA) of disease severity of at least moderate severity (score ≥ 3) as an overall assessment.
5. Subjects with a target lesion which has the following characteristics:

   1. located on the extremities (i.e., arms or legs ) and has an area of ≥25 cm2;
   2. has a minimum plaque erythema of at least moderate severity (PASI grade ≥ 3);
   3. has a minimum plaque scaling severity of at least moderate severity (PASI grade ≥ 3);
   4. has a minimum plaque elevation of at least moderate severity (PASI grade ≥ 3);
6. If females of childbearing potential, the subject must have a negative urine pregnancy test, and must have been using an acceptable form of birth control for at least two months prior to Visit 1/Screening and are willing to continue birth control throughout the study.
7. Subjects must be willing and able to understand and comply with the requirements of the study, apply the assigned investigational product as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study.
8. Subjects must be in good health, as confirmed by medical history and physical exam, and free from any clinically significant disease/condition, other than plaque psoriasis, that might interfere with the study evaluations.
9. Subjects must be willing to limit sun exposure overall. Subjects are prohibited from sunbathing or intentional tanning or intense sun exposure including the use of tanning booths/lights or other artificial UV light sources throughout the study.

Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or planning a pregnancy within the study participation period.
2. Subjects who have a current diagnosis of guttate, pustular, inverse, exfoliative, or erythrodermic psoriasis.
3. Subjects who have a history of psoriasis unresponsive to topical treatments.
4. Subjects who have a history of a disorder that may interfere with the evaluation of plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis, cutaneous lymphoma, etc.).
5. Presence of pigmentation, extensive scarring, or pigmented lesions in the treatment areas, which could interfere with the rating of efficacy parameters.
6. Subjects with unstable medical disorders, life-threatening disease, or current malignancies.
7. Subjects with clinically significant ECG or laboratory abnormalities at Visit 1/Screening (as determined by the Principal Investigator or designee).
8. Subjects who are immunosuppressed.
9. Subjects who have a history of allergy or a known hypersensitivity to any component of the investigational product.
10. Subjects who have been treated with any systemic steroids within the 4 weeks prior to the study entry (intranasal or inhaled corticosteroids are acceptable if kept constant throughout the study, and intra-articular steroid injections are permissible).
11. Subjects who have been treated with systemic or photo antipsoriatic therapies/drugs within 4 weeks prior to study entry including methotrexate, cyclosporine, acitretin and other oral retinoids, broadband or narrowband UVB, PUVA, home or professional tanning lights or other nonprescription UV light sources, photodynamic therapy (PDT), lasers, mycophenalate mofetil (MMF), thioguanine, hydroxyurea, sirolimus, azathioprine, 6-mercaptopurine (6-MP), or etanercept.
12. Subjects who have been treated with biologic therapy other than etanercept within 8 weeks prior to study entry, including adalibumab, infliximab, ustekinumab, golimumab, or rituximab. Vaccines will not be considered an exclusionary biologic treatment.
13. Subjects treated with any other biologic agent not listed here for psoriasis or psoriatic arthritis within 12 weeks.
14. Subjects who have been treated with any topical anti-psoriatic (e.g., salicylic acid, anthralin, tar, etc.,) any topical corticosteroid medications, topical retinoids (e.g., tazarotene, tretinoin), topical Vitamin D analogs (e.g., calcipotriene), topical immunosuppressants (e.g., tacrolimus, pimecrolimus) within 2 weeks prior to study entry.
15. Subjects who have been treated with lithium, antimalarial agents, or quinidine within the 4 weeks prior to study entry.
16. Subjects who have received radiation therapy and/or anti-neoplastic agents, or taken any immunosuppressant medication within 3 months prior to study entry.
17. Subjects who consume excessive amounts of alcohol, abuse drugs, or have any condition that would compromise compliance, in the investigator's opinion, with this protocol.
18. Subjects who have been treated with an investigational drug or investigational device within a period of 30 days prior to study entry, and within 120 days for investigational biologic agent.
19. Subjects who have been previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08-15 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment of Disease Severity (IGA) | 12 weeks
  An assessment of disease severity will be performed at each study visit

SECONDARY OUTCOMES:
Target Lesion Psoriasis Area Severity Index (PASI) | 12 weeks
  Erythema, Scaling and Plaque Elevation of the target lesion will be scored at baseline and at each subsequent study visit.
Body Surface Area (BSA) | 12 weeks
  The % BSA of all treatable psoriatic lesions and regions will be recorded at baseline and at week 12.
Target Lesion Area | 12 weeks
  The target lesion area will be measured at baseline and each-post-baseline visit.
Dermatology Life Quality Index (DLQI) | 12 weeks
  Measured at baseline and week 12

CONTACTS AND LOCATIONS:
Locations (2):
- Dominican Republic (2):
  - Instituto Dermatogical y Cirugia de Piel, San Cristóbal
  - Instituto Dermatologico Blanco Falette, MD, Santo Domingo

IPD SHARING:
Plan to Share IPD: No